CLINICAL TRIAL: NCT03316924
Title: Mecanical Properties of Biomaterials and Biological Integration of Diaphragmatic Prothesis in Infancy
Brief Title: Analysis of in Vitro Biological Reaction of Diaphragmatic Prothesis When Congenital Diaphragmatic Hernia (CDH) Repair
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6834
Record Dates: First submitted 2017-10-17; First posted 2017-10-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-07

CONDITIONS: Congenital Diaphragmatic Repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Foreskin resection — During the pediatric surgery consultation, the doctor will decide between Foreskin resection, orchidopexie or inguinal hernia repair.
  Other Names: orchidopexie; inguinal hernia repair

SUMMARY:
In case of CDH, the incomplete development of a part of the diaphragm allows abdominal viscera to herniate into thorax cavity during fetal development and impaired lung and heart development.

After birth, CDH patients who survived thanks to an active reanimation management undergo diaphragmatic repair. In case of large defect, a patch is needed to complete diaphragmatic closure. Thanks to primary cell culture from foreskin, peritoneal epithelium or cremaster dedicated to incineration investigators want to analyse biological integration of actually used prothesis and others innovations.

ELIGIBILITY:
Inclusion Criteria:

* Minor aged 0 (day of birth) to 14 years
* Patient for whom an indication of posthectomy and / or cure of inguinal hernia and / or testicular ectopy is retained
* Patient whose legal representatives have agreed to the use of operational waste from mesenchymal tissues (foreskin, cremaster and peritoneum) destined for incineration.
* Patient affiliated to a social security scheme

Exclusion Criteria:

- parents don't agree to the use of its operating waste for research purposes

Ages: 0 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children that benefits of a foreskin resection, inguinal hernia repair or orchidopexy
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
cell colonization | samples are processed immediately after sampling
  Study cell colonization
quality of the extracellular matrix | samples are processed immediately after sampling
  Quality of the extracellular matrix produced in vitro in contact with the currently used implant materials compared to biomaterials under development

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle TALON, MD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided